CLINICAL TRIAL: NCT06195813
Title: Effects of Asparagus Capsule Consumption on Blood Sugar and Lipids and Oxidative Stress in Overweight and Obese Participants
Brief Title: Asparagus Capsule Consumption and Blood Sugar and Lipids and Oxidative Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB3-115/2565
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Asparagus Capsule Consumption

STUDY DESIGN:
Intervention Model Description: Participants were randomly divided into 2 groups consisting of 23 asparagus capsules and 21 placebo capsules groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asparagus capsule (Experimental): Participants were randomized to receive an arm. In this arm, participants received asparagus capsule and were asked to consume at 40 mg/kg (1-2 capsule) within 15-30 min after breakfast. Consumption was taken at participants' dwelling.
  Interventions: Dietary Supplement: Asparagus capsule
- Placebo capsule (Placebo Comparator): Participants were randomized to receive an arm. In this arm, participants received placebo capsule and were asked to consume at 40 mg/kg (1-2 capsule) within 15-30 min after breakfast. Consumption was taken at participants' dwelling.
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Asparagus capsule — Asparagus capsule is categorized as dietary supplement.
  Arms: Asparagus capsule
Other: Placebo capsule — Placebo capsule is categorized as other.
  Arms: Placebo capsule

SUMMARY:
Participants were 44 overweight and obese persons, male and female, age 18-59 years. Participants were divided into 2 groups consisting of 23 asparagus capsules and 21 placebo capsules groups. They received health screenings including history taking, mental health questionnaire, and vital signs, height and body weight, body composition, fat distribution measurements and oral glucose tolerance test. Then, a venipuncture was conducted to determine blood glucose, insulin, lipids malondialdehyde and protein carbonyl levels.

DETAILED DESCRIPTION:
The study design was cross-sectional. Participants were 44 overweight and obese persons, male and female, age 18-59 years. Participants were divided into 2 groups consisting of 23 asparagus capsules and 21 placebo capsules groups. They received health screenings including history taking, mental health questionnaire, and vital signs, height and body weight, body composition, fat distribution measurements and oral glucose tolerance test. Then, a venipuncture was conducted to determine blood glucose, insulin, lipids malondialdehyde and protein carbonyl levels. Analysis of covariance was used to analyze parameters between groups and paired t-test was used to analyze parameters intra-group.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged between 18 to 59 years
* Body mass index more than 23 (Asian criteria)
* No history of hypertension, diabetes, cardiovascular disease, respiratory disease, endocrine disease, neuromuscular disease, musculoskeletal disease, liver disease, renal disease, immune disease, infectious disease, or cancer
* No regular intake of dietary supplements, i.e., vitamins, antioxidants
* No regular smokers or alcohol drinkers (>2 times per week)
* Not sportman or regular exerciser (>2 times per week or >150 min per week)
* No food allergy, especially shoot

Exclusion Criteria:

- Current signs or symptoms of infection, i.e., fever, hyperpnea, dyspnea, and palpitations.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Level of body fat | Day 0 and end of 12 weeks
  Level of body fat was measured in percentage unit
Level of fat mass | Day 0 and end of 12 weeks
  Level of fat mass was measured in kilogram unit
Level of fat distribution | Day 0 and end of 12 weeks
  Level of fat distribution was measured by ratio of waist (centimeter) to hip (centimeter)
Concentration of blood glucose | Day 0 and end of 12 weeks
  Concentration of blood glucose was measured in serum in mmol/L unit
Concentration of blood insulin | Day 0 and end of 12 weeks
  Concentration of blood insulin was measured in serum in uU/mL (microunit/milliliter) unit
Concentrations of blood lipids | Day 0 and end of 12 weeks
  Concentrations of total cholesterol, triglyceride, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol were measured in serum in mg/dL unit
Concentration of blood malondialdehyde | Day 0 and end of 12 weeks
  Concentration of blood malondialdehyde was measured in plasma in uM (micromolar) unit
Concentration of blood protein carbonyl | Day 0 and end of 12 weeks
  Concentration of blood protein carbonyl was measured in plasma in nmol/mg protein unit

SECONDARY OUTCOMES:
Concentrations of blood glucose from oral glucose tolerance test | At 0 minute before glucose consumption and at 30, 60, 90, 120 minutes after glucose consumption
  Concentrations of blood glucose were measured before and after glucose consumption at 75 g/100 ml in mg/dL unit

CONTACTS AND LOCATIONS:
Overall Officials: Piyapong Prasertsri, Ph.D., Principal Investigator — Burapha University
Locations (1):
- Faculty of Allied Health Sciences, Burapha University, Mueang, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.